CLINICAL TRIAL: NCT00295035
Title: Phase III Trial of Gemcitabine, Curcumin and Celebrex in Patients With Metastatic Colon Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: tasmc-05-na-05160-ctil
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2006-02

CONDITIONS: Colon Neoplasm
MeSH Terms: conditions — Colonic Neoplasms | interventions — Celecoxib; Curcumin

INTERVENTIONS:
Drug: CELECOXIB
Drug: CURCUMIN

SUMMARY:
Colorectal cancer is a major health concern in the Western world with an estimated lifetime risk of 5-6%. The goal of achieving effective cancer prevention is driven by the prediction that CRC will become the leading cause of death (surpassing heart disease) in this decade, with an estimated 1,000,000 new cases and over 500,000 deaths per year, worldwide. Despite continuing advances in diagnosis and therapy, long-term survival rates have not improved significantly over the last four decades. Nearly 50% of all CRC patients will die of the disease. Preventive strategies offer the best hope, at least until our understanding of the biology of cancer matures to the point where it can be implemented into therapy. The search for new chemopreventive compounds with minimal toxicity raises particular interest in phytochemicals.Curcumin (diferuloylmethane) is a natural compound derived from the rhizome of Curcuma Longa, an East Indian plant, commonly called turmeric. It has been shown to possess potent anti-inflammatory and anti-oxidative properties, for which it has a long history of dietary use as a food additive. Curcumin has also a potent anti-proliferative effects against a variety of cancer cell lines in vitro, which stem from its ability to modulate many intracellular signal transduction pathways. Human phase I-II studies found curcumin to be safe, and indicated no dose-limiting toxicity when taken by mouth at doses up to 10 g/day. This data, together with the dismal therapeutic options available for colon cancer patients, suggest that curcumin warrants investigation in this setting. The present study evaluates gemcitabine in combination with curcumin and celecoxib for patients with colon cancer.

DETAILED DESCRIPTION:
The primary end point of the study is time to tumor progression. The study is designed to detect increase in median time to tumor progression from 2.7 months to 4.0 months, with 80% power at a significance level of 5%. This requires approximately 100 patients. The median time to tumor progression of 2.7 months was found in the Investigational New Drug (IND) treatment program for gemcitabine, which enrolled 3023 patients with locally advanced or metastatic colon cance

ELIGIBILITY:
Inclusion Criteria:

3.1.1 Locally advanced or metastatic adenocarcinoma of the colon confirmed by histology or cytology.

3.1.2 Pateint who are qualified for treatment with gemcitabine 3.1.3 No prior chemotherapy for colon cancer. 3.1.4 Performance status 0-2 (ECOG scale). 3.1.5 Age ≥ 18 y. 3.1.6 Adequate hematologic function (ANC ≥ 1500/mm³, platelet count ≥ 100,000/mm³ ).

3.1.7 Adequate hepatic function (total bilirubin ≤ 2.0xUNL and AST, ALT and AP ≤ 5.0xUNL) 3.1.8 adequate renal function (creatinine ≤ 2.0). 3.1.9 Signed informed consent.

Exclusion Criteria:

3.2.1 A history of treated or active central nervous system involvement by the tumor or active neurological disease.

3.2.2 Prior radiation. Patients with disease outside the irradiation field or documented disease progression of previously irradiated disease are eligible.

3.2.3 Unstable medical condition, including uncontrolled diabetes mellitus or hypertension, active infection, unstable CHF, uncontrolled arrhythmias or unstable coagulation disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-03; Study Completion 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Arie Figer, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center